CLINICAL TRIAL: NCT00661271
Title: Mindfulness-based Stress Reduction for Urban Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00002064; R21AT005209 (NIH)
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Stress, Psychological
Keywords: mindfulness; meditation; urban youth; stress reduction; adolescent; Stress reduction for urban youth
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): 8-week mindfulness-based stress reduction program with one retreat session
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR)
- Healthy Topics (Active Comparator): 8-week health education program with one retreat session - based on a health curriculum developed by McGraw/Hill
  Interventions: Behavioral: Healthy topics

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction (MBSR) — 8 weekly sessions with instruction designed to enhance mindfulness--mindful meditation, mindful yoga, and discussion of mindfulness practice, with one retreat session.
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Healthy topics — 8 week health education program with one retreat session
  Arms: Healthy Topics

SUMMARY:
Our uncontrolled study of mindfulness-based stress reduction (MBSR) for urban youth suggests benefits in mental health and quality of life outcomes. To evaluate further the specific effects of MBSR, we are conducting a small randomized controlled trial of the MBSR program compared with a health education program.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted at two urban clinic sites. HIV-positive youth between the ages of 14 and 22 will be recruited and randomized into either an eight-week (with one retreat session) Mindfulness-Based Stress Reduction (MBSR) course (intervention) or an eight-week (with one retreat session) Healthy Topics (HT) course (active control). Measures of psychological functioning, coping, and life satisfaction will take place at baseline, immediately post-program, and 3-months post program. Medical data, including Cluster of Differentiation 4 (CD4) and viral load counts, will also be collected at the three data collection time points.

ELIGIBILITY:
Inclusion Criteria:

* 14-22 year old youth who receive primary care at the Harriet Lane Clinic or Children's Hospital of Philadelphia.

Exclusion Criteria:

* Significant developmental, behavioral, substance abuse, or psychiatric disorders

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2007-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica M Sibinga, MD, MHS, Principal Investigator — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins, Harriet Lane Clinic, Baltimore, Maryland
  - Children's Hospital of Philadelphia, Adolescent Initiative & Special Immunology Clinic, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Webb L, Perry-Parrish C, Ellen J, Sibinga E. Mindfulness instruction for HIV-infected youth: a randomized controlled trial. AIDS Care. 2018 Jun;30(6):688-695. doi: 10.1080/09540121.2017.1394434. Epub 2017 Oct 25. PMID 29067834
- [Derived] Sibinga EM, Perry-Parrish C, Thorpe K, Mika M, Ellen JM. A small mixed-method RCT of mindfulness instruction for urban youth. Explore (NY). 2014 May-Jun;10(3):180-6. doi: 10.1016/j.explore.2014.02.006. Epub 2014 Feb 25. PMID 24767265

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 96 individuals consented to study participation and 93 were randomized. However, only 72 were able to be contacted for subsequent baseline data collection.
Groups:
- MBSR Program: mindfulness-based stress reduction program
  Mindfulness-based stress reduction (MBSR): 8 weekly sessions with instruction designed to enhance mindfulness--mindful meditation, mindful yoga, and discussion of mindfulness practice, with one retreat session.
- HT Program: Health education program.
  Healthy topics: 8-week health education program with one retreat session
Period: Overall Study
Arm/Group | MBSR Program | HT Program
Started | 48 | 45
Completed | 20 | 20
Not Completed | 28 | 25
Not completed — Lost to Follow-up | 28 | 25

BASELINE CHARACTERISTICS:
Population: 96 participants consented; 93 participants were randomized; 72 participants completed baseline data collection
Groups:
- HT Program: Health education program.
  Healthy topics (HT): 8-week health education program with one retreat session
- Total: Total of all reporting groups
Arm/Group | MBSR Program | HT Program | Total
Number analyzed (Participants) | 38 | 34 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] — All study participants were 14-22 years old; however, 17 participants did not report their exact age. 29 participants contributed age data for the MBSR program arm and 26 participants contributed age data for the HT program arm. Population: All study participants were 14-22 years old; however, 17 participants did not report their exact age: 9 participants in the MBSR arm, 8 participants in the HT arm.
  years
    number analyzed (Participants) | 29 | 26 | 55
    (all) | 18.93 (2.42) | 18.46 (2.20) | 18.71 (2.31)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 8 | 8 | 16
  Between 18 and 65 years | 21 | 18 | 39
  Not Reported | 9 | 8 | 17
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 22 | 16 | 38
  Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 34 | 72

OUTCOME MEASURES:

1. Primary Outcome: Mindful Attention and Awareness Scale (MAAS)
Description: * Mindful Attention and Awareness Scale (MAAS) - measures mindfulness with total score range of 1 - 6, where higher scores indicate greater mindfulness
  * Children's Response Style Questionnaire(CRSQ) - measures coping mechanisms along three subscales: rumination (range: 0-3), distraction (range: 0-3) and problem-solving (range: 0-3), where higher scores on any of the subscales indicates more frequent use of that type of coping mechanism
  * Aggression scale - uses total score to measure aggression with a range of 0-6, where higher scores indicated more aggressive behavior
Time Frame: assessed at Baseline, 3 months follow-up, 4-6 months follow-up; scores at 4-6 month follow-up reported
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- MBSR Program: 8 week mindfulness-based stress reduction program
  Mindfulness-based stress reduction (MBSR): 8 weekly sessions with instruction designed to enhance mindfulness--mindful meditation, mindful yoga, and discussion of mindfulness practice.
- HT Program: Health education group--8 weekly sessions of age-appropriate health topics.
  Healthy topics (HT): 8 week health education program
Arm/Group | MBSR Program | HT Program
Number analyzed (Participants) | 38 | 34
units on a scale
  Mindfulness (MAAS) | 3.79 (0.73) | 3.66 (0.88)
  Problem-Solving Coping (CRSQ) | 1.71 (0.83) | 1.56 (0.77)
  Rumination (CRSQ) | 1.54 (0.82) | 1.18 (0.58)
  Distraction (CRSQ) | 1.46 (0.62) | 1.37 (0.73)
  Aggression | 0.96 (1.30) | 1.44 (1.21)

2. Secondary Outcome: Quality of Life
Description: Life satisfaction was measured with the HIV Quality of Life (QOL) measure, which included three subscales: life satisfaction (range: 1-5), illness burden (range: 1-5) and illness anxiety (range: 1-5). For life satisfaction, higher scores indicated higher satisfaction, and for the other two subscales greater scores indicated more issues with illness burden and illness anxiety.
Time Frame: assessed at Baseline, 3 months follow-up, 4-6 months follow-up; scores at 4-6 month follow-up reported
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBSR Program | HT Program
Number analyzed (Participants) | 38 | 34
units on a scale
  Life Satisfaction | 2.22 (0.74) | 1.63 (0.58)
  Illness Burden | 1.86 (0.72) | 1.63 (0.78)
  Illness Anxiety | 2.38 (0.78) | 2.09 (0.80)

ADVERSE EVENTS:
Groups:
- MBSR Program: mindfulness-based stress reduction program
  Mindfulness-based stress reduction (MBSR): 9 weekly sessions with instruction designed to enhance mindfulness--mindful meditation, mindful yoga, and discussion of mindfulness practice.
- HT Program: Health education program
  Healthy topics: 9 week health education program
Arm/Group | MBSR Program | HT Program
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/34
Other Adverse Events (participants affected / at risk) | 6/38 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBSR Program (N=38) | HT Program (N=34)
Headache (General disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Alteration in personality (Psychiatric disorders) | 1 (1) | 0 (0)
General well being (General disorders) | 1 (1) | 0 (0) — Fight in school

LIMITATIONS AND CAVEATS:
Participant attrition during the study period limited post-intervention data for analysis, although attrition was balanced by study arm, maintaining the balance across study arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No